CLINICAL TRIAL: NCT03323645
Title: Prosthetics Registry and Outcomes in Urology at Duke
Acronym: PROUD
Status: Terminated | Type: Observational
Why Stopped: change of study structure and resource allocation
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00086257
Record Dates: First submitted 2017-10-19; First posted 2017-10-27 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-04

CONDITIONS: Penile Implantation
Keywords: prostate cancer; erectile dysfunction; penile prosthesis
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with penile prostheses

SUMMARY:
To establish the Prosthetics Registry and Outcomes in Urology at Duke (PROUD) which will serve as a retro- and prospective data repository that our team will use to optimize patient satisfaction, lower cost and reduce morbidity associated with penile prosthesis implantation. The study team will collect retrospective data from subjects at Duke University and Duke Raleigh Hospitals who have undergone genitourinary prosthesis implantation from January 1, 1996 onward. Prospective data will only be collected from patients seeking care with Dr. Lentz in Duke Raleigh.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Adult (18 years of age or older)
* Inflatable or semi-rigid penile prosthesis placed

Exclusion Criteria:

- Inability to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men with end-stage erectile dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Development of data repository to capture longitudinal outcomes and satisfaction for subjects who receive penile prostheses. | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aaron C Lentz, MD, Principal Investigator — Duke University
Locations (1):
- Duke Raleigh, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No